CLINICAL TRIAL: NCT03248921
Title: The Impact of Obesity on Postoperative Outcomes Following Cardiac Surgery
Acronym: OPOS
Status: Active, not recruiting | Type: Observational
Sponsor: Cardiovascular Research New Brunswick (Other)
Collaborators: Horizon Health Network (Other); Maritime Heart Centre (Other)
Responsible Party: Principal Investigator, Ansar Hassan, MD, PhD, Principal Investigator, Dalhousie University
Other Study IDs: RS#: 2014-2006
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Cardiac Disease; Cardiovascular Syndromes, Metabolic
MeSH Terms: conditions — Obesity; Heart Diseases; Metabolic Syndrome | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following biological samples have been approved for collection: 4 types of adipose tissue (subcutaneous adipose tissue; epicardial adipose tissue; pericardial adipose tissue; peri-aortic adipose tissue); atrial appendage tissue sample; and 8-10mL blood sample (plasma and serum sample).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High-Fit obese: Cardiac surgery patients will be segregated into the high-fit group based on 6 minute walk test distance and other measures of functional capacity
  Interventions: Procedure: cardiac surgery
- Low-Fit obese: Cardiac surgery patients will be segregated into the low-fit group based on 6 minute walk test distance and other measures of functional capacity
  Interventions: Procedure: cardiac surgery

INTERVENTIONS:
Procedure: cardiac surgery — cardiac surgery including non-emergency, elective coronary artery bypass grafting surgery with or without valve surgery, aortic or mitral valve surgery

SUMMARY:
The purpose of this study is to identify measures of obesity, functional capacity, and specific biomarkers that may be predictive of obesity and post-operative outcomes.

DETAILED DESCRIPTION:
Background: Increasing levels of obesity worldwide have led to a rise in the prevalence of obesity-related complications including cardiovascular disease, diabetes, cancers etc. Health care providers believe that obesity has a negative effect on patients undergoing cardiac surgery, with overweight and obese patients being more likely to experience adverse post-operative outcomes. The body mass index (BMI) is the single most used measure for determining obesity classification in clinical practice, without accounting for a patient's level of cardiopulmonary fitness or muscle mass.

Study Design: Patients between the ages of 18 and 75 years undergoing elective cardiac surgery will be consented to participate in this prospective observational trial. Patients are invited to participate in measures of obesity, functional capacity and exercise capacity assessments, quality of life questionnaires, and blood and tissue sampling for biomarker analysis.

Endpoints: Measures other than BMI that could be predictive of short-term and long-term post-operative outcomes. Outcomes of interest include: prolonged length of ventilation, hospital length of stay and all-cause mortality.

Summary: The results of this trial will potentially identify an improved definition of fitness capacity for obese cardiac surgical patients and biomarkers alone or in combination that could identify the potential for adverse outcomes in patients undergoing cardiac surgery. This study will help clinicians better segregate and treat patients pre-operatively based on fitness levels and associated biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* · Provide informed consent

  * Male or female patients who are > 18 years of age
  * Patients must be scheduled to undergo elective, first-time cardiac surgery during routine scheduling times

Exclusion Criteria:

* Patients who are > 75 years of age
* BMI is less than 18.5 kg/m2 and classified as underweight according to the World Health Organization
* Any non-elective first time cardiac surgery patient (eg. in-house urgent patients; emergent patients)
* Any cardiac patients to undergo re-operation
* Simultaneous participation in another study with an investigational study agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled to undergo elective, first-time cardiac surgery will be considered for eligibility to participate in the study. As well, a patient whose BMI is less than 18.5 kg/m2 and classified as underweight by the World Health Organization will be excluded. Only those patients who are classified as being normal weight range or overweight and/or obese may be considered for eligibility to participate as defined by the study objectives regarding post-operative cardiac surgery outcomes in obese patients. Patients in the normal weight range classification will be included as a baseline control participant cohort. Finally, patients over the age of 75 will be excluded so as to eliminate the role that advanced age may play in affecting functional capacity.
Sampling Method: Non-Probability Sample
Enrollment: 610 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Prolonged Hospitalization | post-operative day (POD) 30
  A length of stay of more than 5 days
Prolonged ventilation > 24 hours | post-operative day (POD) 30
  mechanical ventilation for more than 24 hours of invasive (via endotracheal tube or tracheostomy) and/or noninvasive (facial/nasal interface) methods of delivery

SECONDARY OUTCOMES:
all cause mortality | post-operative day (POD) 30 and 1 year post-op
  Patient death, either in hospital or long-term
non fatal myocardial infarction | post-operative day (POD) 30 and 1 year post-op
  Transmural, Subendocardial infarction
Stroke | post-operative day (POD) 30
  Transient, permanent
Respiratory complications | post-operative day (POD) 30
  Pleural effusion, pneumonia
Prolonged ICU length of stay | post-operative day (POD) 30
  length of stay of more than 48 hours
Re-operation for any cause | post-operative day (POD) 30 and 1 year post-op
  re-operation due to complications, bleeding and/or other reasons
Atrial fibrillation | post-operative day (POD) 30 and 1 year post-op
  post-op occurrence requiring treatment
Post-operative length of stay and disposition on discharge | post-operative day (POD) 30 and 1 year post-op
  home, home with care, transfer to other facility, or expired
Wound infection | post-operative day (POD) 30
  infection of sternum or other incisional access sites

CONTACTS AND LOCATIONS:
Overall Officials: Ansar Hassan, MD, PhD, Principal Investigator — New Brunswick Heart Centre, Department of Cardiac Surgery
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aguiar C, MacLeod J, Yip A, Melville S, Legare JF, Pulinilkunnil T, Kienesberger P, Brunt K, Hassan A. Impact of Obesity on Postoperative Outcomes following cardiac Surgery (The OPOS study): rationale and design of an investigator-initiated prospective study. BMJ Open. 2019 Mar 3;9(3):e023418. doi: 10.1136/bmjopen-2018-023418. PMID 30833313
- [Derived] Sarkar S, Legere S, Haidl I, Marshall J, MacLeod JB, Aguiar C, Lutchmedial S, Hassan A, Brunt KR, Kienesberger P, Pulinilkunnil T, Legare JF. Serum GDF15, a Promising Biomarker in Obese Patients Undergoing Heart Surgery. Front Cardiovasc Med. 2020 Jun 24;7:103. doi: 10.3389/fcvm.2020.00103. eCollection 2020. PMID 32671100
- See also: Related Info — https://impart.team/